CLINICAL TRIAL: NCT02745132
Title: Personalized Medicine in HCV Infection: Cognitive Impairments and Brain Anomalies in Chronic Hepatitis C Infected Individuals. Characterization and Potential Reversibility With Direct Antiviral Agents.
Brief Title: Cognitive Impairments in Chronic Hepatitis C Patients and Potential Reversibility With New Agents (CICHepC)
Acronym: CICHepC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CICHepC-PIE15/00079-JCG; PIE15/00079 (Other Grant/Funding Number: Ministerio de Economía y Competitividad, Spain)
Record Dates: First submitted 2016-04-10; First posted 2016-04-20 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis C
Keywords: Chronic, Cognition Disorders; Neurocognition Disorders; Cognitive Impairments; Diffusion Magnetic Resonance Imaging; MRI functional; Verbal fluency
MeSH Terms: conditions — Hepatitis C; Bronchiolitis Obliterans Syndrome; Cognition Disorders; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive evaluation in HCV patients (Other): Neuropsychological evaluation and Brain MRI
  Intervention: The only intervention to be carried out along the study will consist of complete neuro-psychological tests and MRI studies performed at different times.
  Chronic HCV patients who are going to be treated with new DAAs according to current guidelines will be studied: A neuro-psychological battery of tests and brain MRI studies will be performed at different times before and after the end of the treatment. The participation in the study will not influence neither the indication to treat nor the treatment used.
  Anti-HCV regimens will be used according to clinical practice as indicated into the current guidelines
  Interventions: Other: Neuropsychological evaluation and Brain MRI

INTERVENTIONS:
Other: Neuropsychological evaluation and Brain MRI — This is a prospective study. The only intervention planned will consist of performing neuropsychological tests and cerebral MRI that will be carried out on a single group cohort at different times.
  Notwithstanding, we will record the exposure to DAA to assess any change in neurocognitive function and MRI imaging.
  Anti-HCV regimens will be used according to clinical practice as indicated into the current guidelines (1)
  (1)European Association for Study of Liver. EASL Recommendations on Treatment of Hepatitis C 2015. J Hepatol. 2015 Jul;63(1):199-236. doi: 10.1016/j.jhep.2015.03.025. Epub 2015 Apr 21. PubMed PMID: 25911336.

SUMMARY:
The overall aim of this study is to evaluate the prevalence of cognitive impairments and brain anomalies in Chronic Hepatitis C infected individuals and to investigate likely changes in cognition and brain structure and function after treatment with Direct-acting Antivirals (DAAs).

DETAILED DESCRIPTION:
Design: Prospective interventional study.

Chronic HCV infected patients who are going to initiate a DAA-based antiviral regimen according to clinical practice will be recruited to participate in the study. Patients will be treated according to the current national and international guidelines for the treatment of HCV chronic hepatitis. The participation in the study will not influence neither the indication for de treatment nor the type of treatment prescribed. The only intervention in this study refers to the performance of extraordinary neuro-psychological evaluations and MRI studies at different times along the study.

Patients and methods:

This study will be performed in a cohort of 80 patients with CHC (≤ F3). The number of subjects required to test effects with sufficient power over the entire cortex varies between cortical measures (cortical thickness: N=39, surface area: N=21, volume: N=81; 10mm smoothing, power=0.8, α =0.05). For subcortical regions this number is between 16 and 76 subjects, depending on the region (Liem et al., 2015). Sample size calculations performed for functional magnetic resonance using values of medium Cohen's d effect size of 0.6 and 0.7 yield sample sizes of 88, 66 respectively to achieve 80% power at a significance level of 0.05 (Guo et al., 2012). Therefore, the sample size estimated in this project would yield enough power to detect small and medium effects size.

The following studies will be conducted:

1. - Cognitive assessment: The assessment with widely-used neuropsychological test batteries may yield summary scores for the domains: attention and reaction time (Continuous Performance Test (CPT), working memory (digits forward and backward WAIS-III subtest), information processing speed (digit symbol WAIS-III subtest and Trail making test Part A), verbal fluency (letter FAS and category animals subtest), learning and memory (Rey Auditory 2.- Verbal Learning Test (RAVLT) and Rey Copy Figure(RCF)), motor functioning (Grooved Pegboard) and executive functions (Tower of London, Trail making test Part B and Stroop color-word test).
2. - MRI scanning: Imaging data will be acquired at the neurorradiology section of the Hospital Marques de Valdecilla, on a 3T MRI scanner (Achieva, Philips Medical Systems, Best, The Netherlands) at the Neuroradiology Department of "Marques de Valdecilla" University Hospital. Subjects will undergo a 30 minutes protocol that will include a high resolution T1- weighted image, a 64 directions DWI sequence and A BOLD resting state fMRI sequence.
3. - MRI data analysis: It will involve structural, diffusion and functional MRI analyses. These analyses will be conducted by Neuroimaging Platform at the IDIVAL.

3.1.- Structural MRI: we will use the software FreeSurfer (http://freesurfer.net/) to quantify the volume of subcortical structures (amygdala, hippocampus, thalamus, putamen, globus pallidus, and caudate nucleus) and the area, thickness, and volume of 34 cortical structures (Desikan-Killiany atlas).

3.2.- Diffusion MRI: we will use FSL's TBSS and Probtracx tools http://www.fmrib.ox.ac.uk/fsl/index.html) to compare fractional anisotropy values (a measure based on restricted movement of water molecules) in whole brain voxelwise analysis and identify regions (clusters) where white matter is more disorganized.

Also we will perform fiber tracking and study connectivity between different brain areas.

3.3.- Functional MRI (fMRI): resting state fmri will be used to evaluate regional interactions that occur when non performing and specific task. This analysis will be carried out with using SPM software http://www.fil.ion.ucl.ac.uk/spm/) and the toolbox PRONTO (http://www.mlnl.cs.ucl.ac.uk/pronto ).

ELIGIBILITY:
Inclusion Criteria:

* CHC patients 18-75 years old
* Liver fibrosis ≤ F3 in Fibroscan/liver biopsy
* Naive or previous failure to a treatment
* Accept the study and sign the CI

Exclusion Criteria:

* Does not meet the above criteria
* VIH or other viral coinfection
* Hepatocarcinoma
* Other systemic inflammatory diseases (i.e. RA, etc)
* Neurodegenerative diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Continuous Performance Test (CPT) score | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Cognitive impairment, particularly Attention and reaction time

SECONDARY OUTCOMES:
Changes in Digits forward and backward WAIS-III subtest scores | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Cognitive impairment, particularly Working memory
Changes in Digit symbol WAIS-III subtest score | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Information processing speed
Changes in Trail Making Test (TMT) Parts A & B scores | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Information processing speed
Changes in Letter FAS score | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Verbal fluency
Changes in animal category subtest score | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Verbal fluency
Changes in Rey Auditory Verbal Learning Test (RAVLT) scores | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Learning and memory
Changes in Rey Copy Figure(RCF) scores | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Learning and memory
Changes in Grooved Pegboard score | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Motor functioning
Changes in Tower of London score | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Executive functions
Changes in Stroop color-word test scores | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Neuropsychological test to assess Executive functions
Changes in cortical thickness | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Basal Neuroimaging findings in HCV infected patients and changes after DAA treatment (Assesed through structural, diffusion and functional MRI).
Changes in cortical surface área assessed by MRI | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Basal Neuroimaging findings in HCV infected patients and changes after DAA treatment (Assesed through structural, diffusion and functional MRI).
Changes in cortical surface volumen assessed by MRI | Basal and 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Basal Neuroimaging findings in HCV infected patients and changes after DAA treatment (Assesed through structural, diffusion and functional MRI).
Sustained Viral Response | 3, 6 and 12 months after the end of treatment (Sustained Viral Response)
  Data on efficacy of treatments
Advers events | up to 24 weeks
  Data on safety

CONTACTS AND LOCATIONS:
Overall Officials: Javier Crespo García, MDPhD, Principal Investigator — Head of Gastroenterology and Hepatology at Hospital Universitario Marqués de Valdecilla. Professor at the Universidad de Cantabria; Benedicto Crespo Facorro, MDPhD, Principal Investigator — Head of section Of Psychiatry at University Hospital Marqués de Valdecilla. Proffesor of Psychiatry at Department of Psychiatry, School of Medicine
Locations (1):
- Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrnes V, Miller A, Lowry D, Hill E, Weinstein C, Alsop D, Lenkinski R, Afdhal NH. Effects of anti-viral therapy and HCV clearance on cerebral metabolism and cognition. J Hepatol. 2012 Mar;56(3):549-56. doi: 10.1016/j.jhep.2011.09.015. Epub 2011 Oct 23. PMID 22027578
- [Background] Fletcher NF, Wilson GK, Murray J, Hu K, Lewis A, Reynolds GM, Stamataki Z, Meredith LW, Rowe IA, Luo G, Lopez-Ramirez MA, Baumert TF, Weksler B, Couraud PO, Kim KS, Romero IA, Jopling C, Morgello S, Balfe P, McKeating JA. Hepatitis C virus infects the endothelial cells of the blood-brain barrier. Gastroenterology. 2012 Mar;142(3):634-643.e6. doi: 10.1053/j.gastro.2011.11.028. Epub 2011 Dec 1. PMID 22138189
- [Background] Kraus MR, Schafer A, Teuber G, Porst H, Sprinzl K, Wollschlager S, Keicher C, Scheurlen M. Improvement of neurocognitive function in responders to an antiviral therapy for chronic hepatitis C. Hepatology. 2013 Aug;58(2):497-504. doi: 10.1002/hep.26229. Epub 2013 Jun 24. PMID 23300053
- [Background] Bajaj JS, Forton DM. Cognitive improvement after HCV eradication: Extending the benefits. Hepatology. 2013 Aug;58(2):480-2. doi: 10.1002/hep.26481. Epub 2013 Jun 25. No abstract available. PMID 23696270